CLINICAL TRIAL: NCT07076056
Title: A Randomized, Double-blind, Multi-center, Placebo-controlled, Phase III Trial to Evaluate the Efficacy and Safety of DW1026C1 or DW1026C2 Add-on to Metformin in Patients With Type 2 Diabetes Inadequately Controlled With Metformin and Sitagliptin Combination Therapy
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of DW1026C1 or DW1026C2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW1026-301
Record Dates: First submitted 2025-07-13; First posted 2025-07-21 (Actual); Last update posted 2025-07-21 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- DW1026C1 & DW1026C2 placebo & DW1026S placebo (Experimental)
  Interventions: Drug: DW1026C1
- DW1026C1 placebo & DW1026C2 & DW1026S placebo (Experimental)
  Interventions: Drug: DW1026C2
- DW1026C1 placebo & DW1026C2 placebo & DW1026S (Placebo Comparator)
  Interventions: Drug: DW1026S

INTERVENTIONS:
Drug: DW1026C1 — Sitagliptin 100mg+Empagliflozin 10mg
  Arms: DW1026C1 & DW1026C2 placebo & DW1026S placebo
Drug: DW1026C2 — Sitagliptin 100mg+Empagliflozin 25mg
  Arms: DW1026C1 placebo & DW1026C2 & DW1026S placebo
Drug: DW1026S — Sitagliptin 100mg
  Arms: DW1026C1 placebo & DW1026C2 placebo & DW1026S

SUMMARY:
A Randomized, Double-blind, Multi-center, Placebo-controlled, Phase III Trial to Evaluate the Efficacy and Safety of DW1026C1 or DW1026C2 Add-on to Metformin in Patients With Type 2 Diabetes Inadequately Controlled With Metformin and Sitagliptin Combination Therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with Type2 Diabetes
* 19 ≤ Age ≤ 85
* 7.0% ≤ HbA1c ≤ 10.5%

Exclusion Criteria:

* Patients with a history of acute pancreatitis
* Patients with a history of pre-diabetic coma
* Patients with a history of diagnosis of malignant tumors within 5 years prior to visit 1

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
% change of HbA1c | 24 weeks
  % change of HbA1c in week 24 from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Yeouido St. Mary's Hospital The Catholic University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No